CLINICAL TRIAL: NCT04084132
Title: Early Versus Later Re-valving in Tetralogy of Fallot With Free Pulmonary Regurgitation - Combined Cross-sectional and Prospective, Multi-centre, Randomized, Parallel-group Clinical Trial
Brief Title: Early Versus Later Re-valving in Tetralogy of Fallot With Free Pulmonary Regurgitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lars Soendergaard, Clinical Professor, Consultant MD, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VD-2018-512
Record Dates: First submitted 2019-02-25; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Tetralogy of Fallot; Pulmonary Regurgitation
MeSH Terms: conditions — Tetralogy of Fallot; Pulmonary Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early re-valving (Experimental): 60 patients who are assigned to early re-valving undergo pulmonary valve replacement within 3 months from randomization.
  Interventions: Procedure: Pulmonary valve replacement
- Later re-valving (Experimental): 60 patients who are assigned to later re-valving undergo pulmonary valve replacement when the current European guideline criteria are met.
  Interventions: Procedure: Pulmonary valve replacement

INTERVENTIONS:
Procedure: Pulmonary valve replacement — Surgical implantation of an adult-sized (≥ 18 mm) homograft or Contegra graft as right ventricle-to-pulmonary artery conduit under cardiopulmonary bypass through a sternotomy.

SUMMARY:
Tetralogy of Fallot (ToF) is a congenital heart defect with four major features including right ventricular outflow tract obstruction. About 25 children are born with this condition in Denmark every year. Corrective surgery is usually performed within the first year. In 50 % of patients, enlargement with a patch is necessary to achieve relief of the outflow tract obstruction. This however results in severe pulmonary regurgitation, which eventually leads to volume overload, right ventricular dysfunction and arrhythmia. To avoid these late complications, pulmonary valve replacement with a prosthesis if performed when patients meet the current guideline criteria. Most patients meet the guideline criteria for revalving when they are between 20 and 30 years of age. The current guidelines however, are based solely on retrospective studies and novel research reveals that in more than 50 % of patients who are treated according to current practice, right ventricular volumes and function as well as exercise capacity and burden of arrhythmia do not normalize or improve. 500 patients with ToF will be enrolled in a multicentre, cross-sectional study, which will yield information about the long-term outcomes after initial repair of ToF, as well as suggestions about the optimal timing for re-valving. Among patients included in the cross-sectional study, 120 patients with free pulmonary regurgitation, will be randomized evenly for early or later re-valving with at least 10-years of follow-up, for evaluation of long-term efficacy and safety of early re-valving.

ELIGIBILITY:
Inclusion Criteria:

1. ToF with pulmonary stenosis repaired with a TAP within the first two years of life.
2. RVOT anatomy is suitable for implantation of an adult sized conduit ( 18 mm homograft or Contegra graft) as assessed by MRI.

Exclusion Criteria:

1. ToF with pulmonary atresia, ToF with common atrioventricular canal, ToF with absent pulmonary valve syndrome, major aortopulmonary collateral arteries and other significant associated anomalies.
2. Palliation with a shunt (Blalock-Taussig or central) at any time.
3. The patient is symptomatic.
4. Sustained supraventricular or ventricular arrhythmia.
5. RVEDVi > 140 mL/m2 as assessed by MRI (appendix 1).
6. RVESVi > 60 mL/m2 as assessed by MRI.
7. RVEF < 50 % as assessed by MRI.
8. Moderate or severe tricuspid regurgitation as assessed by echocardiography or MRI.
9. Significant residual lesions requiring intervention (e.g. ventricular septal defect, aortic regurgitation, branch pulmonary artery stenosis).
10. Co-morbidity preventing exercise testing (e.g. genetics, neuro-cognitive dysfunction, physical disability).
11. Contraindication for MRI (e.g. permanent pacemaker, intra-cardiac defibrillator, intracranial ferro-magnetic device).
12. Pregnancy at time of inclusion.
13. Age < 12 or unable to comply with instructions given during MRI or exercise testing.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean right ventricular end-diastolic volume indexed to body surface area | 3 years after randomization
  Right ventricular end-diastolic volume (mL) indexed by body surface area (m2) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Higher right ventricular end-diastolic volumes are considered a worse outcome.
Rate of deceased patients (all-cause mortality) and total number of patients | 3 years after randomization
  The rate of deceased patients (irrespective of the cause of death) and total number of patients will be calculated for both the early and later re-valving group and analysis of statistical significance of the difference between the groups will be performed.

SECONDARY OUTCOMES:
Right ventricular end-systolic volume indexed to body surface area | Assessed once every year for 10 years after randomization
  Right ventricular end-systolic volume (mL) indexed by body surface area (m2) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Higher right ventricular end-systolic volumes are considered a worse outcome.
Right ventricular ejection fraction | Assessed once every year for 10 years after randomization
  Right ventricular ejection fraction (%) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Lower right ventricular ejection fraction are considered a worse outcome.
Left ventricular end-diastolic volume indexed to body surface area | Assessed once every year for 10 years after randomization
  Left ventricular end-diastolic volume (mL) indexed by body surface area (m2) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Higher left ventricular end-diastolic volumes are considered a worse outcome.
Left ventricular end-systolic volume indexed to body surface area | Assessed once every year for 10 years after randomization
  Left ventricular end-diastolic volume (mL) indexed by body surface area (m2) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Higher left ventricular end-systolic volumes are considered a worse outcome.
Left ventricular ejection fraction | Assessed once every year for 10 years after randomization
  Left ventricular ejection fraction (%) will be assessed in both the early re-valving group and later re-valving group for calculation of the mean in each group and analysis of statistical significance of the difference will be performed. Lower left ventricular ejection fraction are considered a worse outcome.
Rate of patients with procedure-related bleeding and total number of patients | 30 days after surgery
  The rate of patients with bleeding classified as minor, major and life-threatening bleeding (BARC classification) related to the re-valving procedure and the total number of patients will be calculated in both the early and later re-valving group and the difference between the groups will be analyzed for statistical significance.
Rate of patients with procedure-related acute kidney injury and total number of patients. | 30 days after surgery
  The rate of acute kidney injury categorized as stage one, two and three (KDIGO classification) and the total number of patients will be calculated in both the early and later re-valving group and the difference will be analyzed for statistical significance.
Composite-rate of all-cause mortality and disabling stroke | Assessed once every year for 10 years after randomization
  The rate of patients who decease due to cardiovascular causes and patients who suffer from a disabling stroke after the time of randomization will be calculated for both the early and later re-valving group and the difference will be analyzed for statistical significance
Rate of patients deceased due to cardiovascular causes and total number of patients | Assessed once every year for 10 years after randomization
  The rate of patients who decease due to a cardiovascular cause and the total number of patients will be calculated in both the early and later re-valving group and the difference will be analyzed for statistical significance
Composite-rate of patients who suffer from disabling strokes or transient ischemic attacks | Assessed once every year for 10 years after randomization
  The rate of patients who suffer from a disabling stroke og transient ischemic attack after the time of randomization will be calculated in both the early and later re-valving group and the difference will be analyzed for statistical significance
Mean New York Heart Association class | Assessed once every year for 10 years after randomization
  The mean New York Heart Association Class categorized as 1-4 will be assessed in both the early and later re-valving group and the difference will be analyzed for statistical significance. Higher mean values are considered a worse outcome.
Mean health-associated quality of life (adults) | Assessed once every year for 10 years after randomization
  The mean health-asssociated quality of life will be assessed in both the early and later revalving group and the difference will be analyzed for statistical significance. EQ-5D-3L will be used for assessment. The questionnaires are available in Danish. Higher values are considered better outcomes.
Mean health-associated quality of life (children) | Assessed once every year for 10 years after randomization
  The mean health-associated quality of life will be assessed in both the early and later re-valving group and the difference will be analyzed for statistical significance. EQ-5D-Y will be used for assessment. The questionnaires are available in Danish. Higher values are considered better outcomes.
Rate of patients with new sustained supraventricular or ventricular arrhythmia and the total number of patients | Assessed once every year for 10 years after randomization
  The rate of patients with new supraventricular or ventricular arrhythmia and the total number of patients will be calculated for both the early and later re-valving group and the difference will be analyzed for statistical significance.
Mean peak oxygen consumption during cardiopulmonary exercise testing | Assessed once every year for 10 years after randomization
  The mean peak oxygen consumption (VO2/min) indexed to body weight (kg) will be assessed for patients in both the early and later re-valving group and the difference in means will be analyzed for statistical significance. Higher mean values are considered a better outcomes.
Median time until structural valve deterioration in patients who are re-valved during the study | Assessed once every year for 10 years after randomization
  The median time until structural valve deterioration defined as time until need for valve replacement in patients who are revalved during the study will be calculated.
Rate of patients who are re-valved during the course of the study and suffer from endocarditis and the total number of patients who are revalved during the study | Assessed once every year for 10 years after randomization
  The rate of patients who suffer from endocarditis after re-valving during the course of the study and the total number of patients who are revalved during the study will be calculated
Rate of patients who are re-valved during the course of the study and suffer from prosthetic valve thrombosis and the total number of patients who are revalved during the study | Assessed once every year for 10 years after randomization
  The rate of patients who suffer from prosthetic valve thrombosis after re-valving during the course of the study and the total number of patients who are revalved during the study will be calculated
Mean number of contacts to the health system | Assessed once every year for 10 years after randomization
  The mean number of contacts to the health system defined as composite of hospital admissions, outpatient contacts and contacts to the general practitioner will be calculated in both the early and later re-valving group and the difference will be analyzed for statistical significance
Mean number of children for female patients | Assessed once every year for 10 years after randomization
  The mean number of children will be assessed for female patient in both the early and later re-valving group and the difference will be analyzed for statistical significance

CONTACTS AND LOCATIONS:
Overall Officials: Lars Søndergaard, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark; Morten H Smerup, MD, PhD, Study Chair — Rigshospitalet, Denmark; Dorte G Nielsen, MD, PhD, Study Chair — Aarhus University Hospital; Kim Munk, MD, PhD, Study Chair — Aarhus University Hospital; Henrik Nissen, MD, PhD, Study Chair — Odense University Hospital; Helle Andersen, MD, Study Chair — Odense University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT04084132/Prot_SAP_000.pdf